CLINICAL TRIAL: NCT07199491
Title: Testing a Multilevel, Culturally Appropriate Lifestyle Intervention For Hispanic Patients With Metabolic-dysfunction Associated Steatotic Liver DiseaseTesting a Multilevel, Culturally Appropriate Lifestyle Intervention For Hispanic Patients With Metabolic-dysfunction Associated Steatotic Liver Disease
Brief Title: Testing a Multilevel, Culturally Appropriate Lifestyle Intervention For Hispanic Patients With Metabolic-dysfunction Associated Steatotic Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Natalia Heredia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-25-0539; K01MD019149 (NIH)
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metabolic-dysfunction Associated Liver Disease (MASLD)
Keywords: weight loss; alcohol consumption; Diabetes Prevention Program (DPP)
MeSH Terms: conditions — Weight Loss; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Liver/Hígado Sano program (Experimental)
  Interventions: Behavioral: Healthy Liver/Hígado Sano program
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Healthy Liver/Hígado Sano program — Participants will attend weekly classes over the 6-month period. This consists of 16 core sessions delivered in the first 6 months (weekly, but with flexibility to skip weeks as necessary due to holidays, etc). The sessions are 30-60 minutes long, conducted in a group setting, with a CDC-certified Lifestyle Coach facilitating the sessions.
  Arms: Healthy Liver/Hígado Sano program
Behavioral: Usual Care — participants will first complete a 30- to 45-minute questionnaire that will cover topics such as physical activity, diet, alcohol use, and stress.Participants will then be asked to wear an accelerometer for 7 days and complete a log to identify when it was worn and removed each day.Height and weight will also be measured and a Fibroscan® assessment (to measure amount of fat and scar tissue in the liver), as well as blood work to monitor the liver enzymes will be done
  Arms: Usual Care

SUMMARY:
The purpose of this study is to understand if a behavioral lifestyle intervention called the Healthy Liver/Hígado Sano program can help Hispanic/Latino patients with metabolic dysfunction associated steatotic liver disease (MASLD), also known as non-alcoholic fatty liver disease (NAFLD), lose weight and improve their liver health

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic/Latino
* Have been diagnosed with MASLD
* Able to speak English or Spanish
* Have access to internet, either on their phone, at home or at some other location convenient to the participant
* Have a family member willing to attend all sessions

Exclusion Criteria:

* Does not have a working telephone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participants recruited | Baseline
  Recruitment will be assessed to be feasible if ≥65% of eligible participants enroll in the study
Number of participants that completed the study | 6 months
Number of participants that completed the study | 12 months
Number of participants that adhered to the protocol | 6 months
Number of participants that adhered to the protocol | 12 months
Participant satisfaction as assessed by the Client Satisfaction Questionnaire (CSQ-8) | 6 months
  The CSQ-8 is an 8-item self-report instrument assessing satisfaction with services received. Each item is rated on a 4-point Likert scale (1 = least satisfied, 4 = most satisfied). Item scores are summed to produce a total score ranging from 8 to 32, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Change in physical activity using the self-reported International Physical Activity Questionnaire(IPAQ) | Baseline, 6 months, 12 months
  This is a 27 item questionnaire assessing the frequency (days per week) and duration (minutes per day) of physical activities across four domains: work, transportation, household/gardening, and leisure-time, as well as time spent sitting. Physical activity scores are calculated in metabolic equivalent task minutes per week (MET-minutes/week) by multiplying activity intensity (Walking = 3.3 METs, Moderate = 4.0 METs, Vigorous = 8.0 METs) × duration × frequency within each domain. Total physical activity is obtained by summing across all domains, and respondents are classified into Low, Moderate, or High activity categories according to standardized IPAQ scoring guidelines.
Change in physical activity as assessed by the Actigraph GT9X accelerometers | Baseline, 6 months, 12 months
Change in diet as assessed by the National Cancer Institute's Family Life, Activity, Sun, Health, and Eating (FLASHE) dietary screener self reported questionnaire | Baseline, 6 months, 12 months
  This is a 27-item questionnaire that captures past 7-day consumption of fast and junk foods, sugary foods/desserts, fruits and vegetables, and sugar-sweetened beverages. Each item is scored based on reported frequency (ranging from "Never" to "2 or more times per day"). For each food category, responses are converted to frequency per day. Higher frequencies indicate greater reported intake of that food category
Change in weight | Baseline, 6 months, 12 months
Change in Liver steatosis (fatty liver disease) and/or stiffness assessed using the Fibroscan data | Baseline, 6 months, 12 months
Change in liver steatosis (fatty liver disease) and/or stiffness using liver enzyme information using blood draws | Baseline, 6 months, 12 months
Change in fasting glucose levels | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Heredia, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No